CLINICAL TRIAL: NCT00649922
Title: Assessment of the Effect of Adalimumab on Response to Influenza Virus and Pneumococcal Vaccines in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Lawrence McNamee, Sr. Clinical Research Manager, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M03-600
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Vaccines with adalimumab dosing
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double Blind (Placebo Comparator)
  Interventions: Biological: adalimumab; Biological: placebo
- Open Label (Experimental)
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — 80 mg adalimumab (2 injections) day 1; 40 mg (1 injection) Day 15 and Day 29
  Other Names: ABT-D2E7; Humira
  Arms: Double Blind
Biological: placebo — 2 injections Day 1, 1 injection Days 15 and 29
  Arms: Double Blind
Biological: adalimumab — 40 mg adalimumab every other week
  Other Names: ABT-D2E7; Humira
  Arms: Open Label

SUMMARY:
To evaluate the immunogeneicity of the Influenza virus and standard 23-valent pneumococcal virus in subject with RA receiving adalimumab or placebo

ELIGIBILITY:
Inclusion Criteria:

* Male/Females at least 20 years of age.
* Females post-menopausal for at least 1 year, surgically sterile, or practicing acceptable methods of birth control.
* Females have a negative pregnancy test at screening.
* Diagnosis of RA and met ACR criteria.
* Must discontinue any TNF at least 2 months prior to baseline.
* In condition of general good health.

Exclusion Criteria:

* History of significant sensitivity to any drug; clinically significant drug or alcohol abuse within the past year; active infection with Listeria or TB; lymphoma or leukemia; sickle-cell disease, splenectomy, other malignancy within 5 years with the exception of successfully treated non-metastatic basal cell or squamous cell carcinoma of skin or localized carcinoma in situ of the cervix.
* History of current acute inflammatory joint disease.
* Use of TAMIFLU or Symmetrel within 3 months of study drug administration.
* Recent (3 month) history of influenza or pneumococcal bacterial infection.
* Known positive human immunodeficiency virus (HIV) status.
* Positive hepatitis B or hepatitis C virus.
* Positive PPD >5 mm.
* Chest x-ray with calcified granulomas and/or pleural scarring or significant abnormalities.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2003-10; Primary Completion 2004-12 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Blood samples for Influenza A & B antibody Assay | Baseline (Day 1), Day 36 or premature discontinuation
Blood Samples for Pneumococcal Antibody Assay | Baseline (Day 1), Day 36 or premature discontinuation

SECONDARY OUTCOMES:
Laboratory assessments | Screening, Week 15, Day 36, Month 3 and Month 6
Vitals signs | Screening - Month 6
Adverse events | Screening - Month 6

REFERENCES:
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778